CLINICAL TRIAL: NCT04078997
Title: Pneumococcal Conjugate Vaccine 13 (PCV13) Schedule Change From 3+0 to 2+1 to Accelerate Reduction in Pneumococcal Vaccine Serotype Carriage in Blantyre, Malawi: an Effectiveness Study
Brief Title: An Evaluation of PCV13 Vaccine Schedules, Comparing Impact of 2+1 vs 3+0 on Pneumococcal Carriage in Blantyre, Malawi
Acronym: PAVE
Status: Completed | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); Ministry of Health, Malawi (Other Government); Blantyre District Health Office (Unknown); UNICEF (Other); World Health Organization (Other); University College, London (Other); Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 5270; OPP1208803 (Other Grant/Funding Number: The Bill & Melinda Gates Foundation)
Record Dates: First submitted 2019-08-28; First posted 2019-09-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-07

CONDITIONS: 13-valent Pneumococcal Vaccine; Streptococcus Pneumoniae
Keywords: Pneumococcal carriage; Pneumococcal conjugate vaccine; Vaccine schedule; Evaluation; Children; Herd immunity; Malawi

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Frozen samples with isolated DNA will be retained, confirming to requirements of the local research ethics committee.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- PCV13-vaccinated,15-24 months of age: Recruitment for carriage surveillance (primary endpoint) will take place at randomly selected households within each of the catchment areas (zones) of the 20 selected health centers.
  Sampling: Random sampling from populations will occur preferentially around the health centers and not from the population on the zonal interfaces. Researchers will designate two geographic sampling areas within each zone around each health center that allows a buffer against zonal borders. If the recruitment target within first sampling area is not met, sampling will move into the second area.
  Interventions: Other: nasopharyngeal swab
- PCV13-vaccinated, 5-10 years of age: Six schools will be selected: three located centrally in each of the 3+0 zones, and three in the 2+1 zones.
  Sampling: Children will be randomly chosen and recruited from each school. NP swab collection will occur during two surveys, starting 21 and 34 months after the switch to 2+11.
  Mapping analysis from our current surveillance activities shows good clustering of recruited children living around the school, suggesting limited movement and thus low risk of contamination between zones with different vaccination schedules.
  Interventions: Other: nasopharyngeal swab
- PCV13-unvaccinated HIV-infected adults on ART 18 - 40 years of: Adults will be recruited from the Queen Elizabeth Central Hospital (QECH), Lighthouse ART clinic in Blantyre.
  Sampling: Mapping analysis from current surveillance activities shows good distribution throughout the Blantyre area, suggesting it is possible to achieve balance between those adults residing in 2+1 vs 3+0 areas. Sample collection will be on a rolling basis throughout the study period, starting 18 months after switch to 2+1.
  Interventions: Other: nasopharyngeal swab
- PCV13-vaccinated, 9 months of age: Recruitment will take place at vaccination centers.
  Sampling: A convenience sample of NP swabs will be collected at the 9-month (measles-1) visit. Sample collection will occur 9 months after the switch to 2+1 schedule.
  Interventions: Other: nasopharyngeal swab

INTERVENTIONS:
Other: nasopharyngeal swab — A nasopharyngeal swab will be collected from consenting individuals by inserting a commercially-available dacron swab to the nasopharynx, gently rotating before removing.

SUMMARY:
Pneumococcal conjugate vaccines (PCV) have been shown to be effective against invasive pneumococcal disease (IPD; including pneumococcal meningitis and sepsis) and all-cause mortality among young children when introduced into infant expanded programs on immunization (EPI). Colonization of the nasopharynx by Streptococcus pneumoniae is a necessary prerequisite to pneumococcal disease. Critically important to the population impact of PCV is therefore reducing vaccine serotype (VT) carriage prevalence, and therefore reducing both disease and onward transmission to vulnerable individuals. Thus, as well as protecting the vaccinated individual (direct protection), PCV confers indirect protection (herd immunity) to unvaccinated populations and to vaccinated individuals who have insufficient protective immunity.

While the ability of PCVs to induce herd immunity has been strong enough to control pneumococcal carriage in industrialized countries, such benefits have not been as marked in low-income countries. Carriage surveillance in Blantyre, Malawi from 4 to 7 years post-vaccine implementation shows persistent VT carriage. With the exception of South Africa, most sub-Saharan African countries, including Malawi, have introduced PCV using a 3+0 schedule. Whether the WHO-approved 2+1 schedule will maximize vaccine-induced protection has been identified as a research gap by the WHO. In this context, the Malawian Ministry of Health (MoH) and the National Immunizations Technical Advisory Committee (NITAG) are seeking evidence of adequate superiority of a 2+1 schedule to inform a change to the current Malawi EPI schedule.

HYPOTHESIS: Prolonging the period of vaccine-induced protection with a booster vaccine dose at 9 months will extend the period of low VT carriage, hence providing longer direct vaccine-induced protection as well as boosting the indirect herd immunity effect.

METHOD: The MoH will implement an evaluation, comparing a 2+1 to the current 3+0 PCV13 vaccine schedule in Blantyre District. This will use a pragmatic health centre-based randomization protocol, implemented within the scope of the EPI programme. This MoH-led change will be evaluated in partnership with the Malawi Liverpool Wellcome Trust Clinical Research Programme. Community carriage surveillance will be undertaken at 15 and 33 months after the introduction of the 2+1 schedule.

The primary endpoint will be VT carriage prevalence among children 15-24 months of age 36 months after schedule change. Other targeted study groups will include children aged 5-10 years who have received PCV13 on a 3+0 schedule, children aged 9 months who have received PCV13 in either a 3+0 or a 2+0 schedule, and HIV-infected adults aged 18-40 years receiving ART and PCV13-unvaccinated.

EXPECTED FINDINGS: Data will inform NITAG decisions on national vaccine policy, with implications at a national, regional and global level.

DETAILED DESCRIPTION:
STUDY TYPE: Pragmatic health center-based evaluation to compare effectiveness of a MoH-mandated structured PCV13 schedule change from 3+0 to 2+1 dosing in a high disease burden setting in Malawi PROBLEM: Streptococcus pneumoniae is a leading cause of childhood pneumonia, meningitis, and bacteremia in sub-Saharan Africa. Pneumococcal conjugate vaccines (PCV) the commonest pneumococcal serotypes have been shown to be effective against pneumococcal meningitis and sepsis, so-called invasive pneumococcal disease (IPD), pneumonia, and all-cause mortality among young children when introduced into infant expanded programs on immunization (EPI). Colonization of the nasopharynx by Streptococcus pneumoniae is a necessary prerequisite to pneumococcal disease. Critically important to the population impact of PCV is therefore reducing vaccine serotype (VT) carriage prevalence, and therefore reducing both disease and onward transmission to vulnerable individuals. Thus, as well as protecting the vaccinated individual (direct protection), PCV confers indirect protection (herd immunity) to unvaccinated populations and to vaccinated individuals who have insufficient protective immunity.

While the ability of PCVs to induce herd immunity has been strong enough to control pneumococcal carriage and disease in industrialized countries, such benefits have not been as marked in low-income countries. In Malawi, the introduction of the PCV13 achieved an approximate 70% reduction in IPD among vaccinated children, and an estimated 35% fall in all-cause mortality among vaccinated children. However, carriage surveillance 4 to 7 years post-vaccine implementation shows persistent VT carriage. Data suggests that most of the vaccine's direct benefit occurs in the first 12 months of life, further suggesting that vaccine-induced protection against pneumococcal disease and colonization wanes rapidly under the current 3+0 schedule. With the exception of South Africa, most sub-Saharan African countries, including Malawi, have introduced PCV using a 3+0 schedule (doses at 6, 10, and 14 weeks of age). Whether the 2+1 schedule (6, 10 weeks and 9 months of age) will maximize vaccine-induced protection has been identified as a research gap by the WHO. There is a dearth of head-to-head studies directly comparing these two schedules. In this context, the Malawian Ministry of Health (MoH) and the National Immunizations Technical Advisory Committee (NITAG) are seeking evidence of adequate superiority of a 2+1 schedule to inform a change to the current Malawi EPI schedule.

HYPOTHESIS: Prolonging the period of vaccine-induced protection with a booster vaccine dose at 9 months will extend the period of low VT carriage, hence providing longer direct vaccine-induced protection as well as boosting the indirect herd immunity effect.

METHOD: The MoH will implement a 2+1 PCV13 vaccine schedule change in Blantyre District. A comparison with the ongoing 3+0 schedule will use a pragmatic health centre-based randomization protocol, with 10 centres continuing with the current 3+0 and 10 implementing the WHO-approved 2+1 schedule. This change will be implemented within the scope of the EPI, subjected to EPI standard procedures for delivery, monitoring, and assessment. This MoH-led change will be evaluated as part of a longstanding partnership with the Malawi Liverpool Wellcome Trust Clinical Research Programme. Researchers will undertake two population based pneumococcal carriage surveys in these 20 health centre catchment areas, at 15 and 33 months after the introduction of the 2+1 schedule.

PRIMARY OUTCOME: VT carriage prevalence among children 15-24 months of age 36 months after schedule change.

SECONDARY OUTCOMES: VT carriage prevalence among children 5-10 years old, among HIV infected adults 18-40 years, add among children 9 months old. Others include prevalence of multiple serotype carriage, and completeness of 3 doses PCV13.

POPULATION: Children who are aged 15-24 months, residents of Blantyre District, and who have received PCV13 in either a 3+0 or a 2+1 schedule (recruited from households); Children aged 5-10 years who have received PCV13 on a 3+0 schedule (recruited from schools); children aged 9 months, who have received PCV13 in either a 3+0 or a 2+0 schedule (recruited from health centres at routine 9-month visit); HIV-infected adults aged 18-40 years receiving ART and PCV13-unvaccinated (recruited from the Queen Elizabeth Central Hospital (QECH) HIV/ART Clinic) EXPECTED FINDINGS: Data will inform NITAG decisions on national vaccine policy, with implications at a national, regional and global level. Results will be disseminated through peer-reviewed publications, scientific conferences, and other relevant stakeholder and policymakers' meetings. This work will strengthen collaboration between relevant government and academic institutions, provide research training for MoH staff and early-career researchers.

ELIGIBILITY:
INCLUSION CRITERIA

PCV13-vaccinated children, 15-24 months of age (schedule 2+1 or 3+1):

* Aged between 15-24 month
* Permanent resident in Blantyre District
* Parent/legal guardian consent for the child to have a NP swab taken
* Evidence of having received a full schedule of PCV13 vaccination recorded in the health passport and which schedule given

PCV13-vaccinated children, 9 months of age (schedule 2+0 or 3+0):

* Aged 9 months
* Permanent resident in Blantyre District
* Parent/legal guardian consent for the child to have a NP swab taken
* Evidence of having received either a full 3+0 schedule or both primary doses (at approximately 6 and 14 weeks of age) of the 2+1 schedule of PCV13 vaccination recorded in the health passport

PCV13-vaccinated children, 5-10 years of age (schedule 3+0):

* Aged between 5-10 years
* Parent/legal guardian consent for the child to have a NP swab taken
* If the child is ≥8 years old, child assent to have a NP swab taken
* Either verbal or documented evidence of having received primary immunization with PCV

PCV13-unvaccinated HIV-infected adults on ART 18 - 40 years of age:

• Aged 18-40 years

EXCLUSION CRITERIA:

For all participants:

* Current TB treatment
* Pneumonia hospitalization <14 days before study enrolment
* Terminal illness

For Children:

* No parental/legal guardian consent
* No child assent (children aged >8 years old)
* Having received antibiotic treatment <14 days before study enrolment

For Adults:

* Unable or unwilling to provide consent
* Prior vaccination with pneumococcal vaccine

Ages: 15 Months to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: PCV13-vaccinated,15-24 months of age: Recruitment at randomly selected households within each of the catchment areas (zones) of the 20 selected health centers.
  PCV13-vaccinated, 9 months of age: Recruitment will take place at MoH EPI vaccination centers.
  PCV13-vaccinated, 5-10 years of age: Recruitment from six selected six schools: three located centrally in each of the 3+0 zones, and three in the 2+1 zones.
  PCV13-unvaccinated HIV-infected adults on ART 18 - 40 years old: Recruitment from the Queen Elizabeth Central Hospital (QECH), Lighthouse ART clinic in Blantyre.
Sampling Method: Probability Sample
Enrollment: 3507 (Actual)
Dates: Start 2019-07-21 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Vaccine-type pneumococcal carriage prevalence among children 15-24 months old | 36 months after 2+1 vaccine schedule implementation

SECONDARY OUTCOMES:
Vaccine-type pneumococcal carriage prevalence among children 5-10 years old | 36 months after 2+1 vaccine schedule implementation
Vaccine-type pneumococcal carriage prevalence among HIV infected adults 18-40 years old | 36 months after 2+1 vaccine schedule implementation
Vaccine-type pneumococcal carriage prevalence among children 9 months old | 9 months after 2+1 vaccine schedule implementation
Prevalence of multiple pneumococcal serotype carriage | 36 months after 2+1 vaccine schedule implementation
Proportion of children receiving a full 3-dose PCV13 vaccination schedule | 36 months after 2+1 vaccine schedule implementation

CONTACTS AND LOCATIONS:
Overall Officials: Robert Heyderman, PhD, Principal Investigator — University College, London; Stephen Gordon, PhD, Study Chair — Malawi-Liverpool-Wellcome Trust Clinical Research Programme
Locations (1):
- Malawi-Liverpool-Wellcome Research Programme, Blantyre, Chichiri, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roessler W, Steinbach P, Nicolai H, Hofstaedter F, Wieland WF. Effects of high-energy shock waves on the viable human kidney. Urol Res. 1993;21(4):273-7. doi: 10.1007/BF00307710. PMID 8212416
- [Derived] Swarthout TD, Ibarz-Pavon A, Kawalazira G, Sinjani G, Chirombo J, Gori A, Chalusa P, Bonomali F, Nyirenda R, Bulla E, Brown C, Msefula J, Banda M, Kachala J, Mwansambo C, Henrion MY, Gordon SB, French N, Heyderman RS. A pragmatic health centre-based evaluation comparing the effectiveness of a PCV13 schedule change from 3+0 to 2+1 in a high pneumococcal carriage and disease burden setting in Malawi: a study protocol. BMJ Open. 2021 Jun 17;11(6):e050312. doi: 10.1136/bmjopen-2021-050312. PMID 34140345